CLINICAL TRIAL: NCT00491699
Title: A Phase 1 Dose Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of XL999 Administered Intravenously to Subjects With Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: Safety Study of XL999 in Adults With Non-Small-Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped due to safety concerns
Sponsor: Symphony Evolution, Inc. (Industry)
Responsible Party: Charles W. Finn, PhD, President and CEO, Symphony Evolution, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL999-002
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: XL999 — XL999 will be administered as a once-weekly 4 hour IV infusion as a single agent. The first cohort will be dosed at 0.4 mg/kg IV once weekly. The maximum dose cohort will not exceed 1.6 mg/kg IV once weekly. Ten subjects are planned for each dosing cohort, with dose escalation dependent on safety and available PK data from prior cohorts

SUMMARY:
The purpose of this study is to determine the safest dose of XL999 and how well subjects with Non-Small-Cell Lung Cancer tolerate XL999. XL999 is a small molecule inhibitor of multiple kinases including VEGFR, PDGFR, FGFR, FLT-3, and Src, which are involved in tumor cell growth, formation of new blood vessels (angiogenesis), and metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a confirmed histological diagnosis of NSCLC.
2. The subject has previously been treated with a platinum- or taxane-containing regimen.
3. The subject has stage IIIB NSCLC with malignant effusion, stage IV or recurrent NSCLC that is not amenable to curative therapy (either surgery or radiation therapy).
4. The subject is at least 18 years old.
5. The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
6. The subject has a life expectancy of ≥3 months.
7. The subject has adequate organ and marrow function.
8. The subject has cardiac-specific enzyme levels (creatine phosphokinase [CPK] total, CPK-MB, and troponin) below the institution's ULN.
9. The subject is capable of understanding the protocol and has signed the informed consent document.
10. Sexually active subjects (male and female) must use medically accepted methods of contraception during the entire course of the study.
11. Female subjects of childbearing potential must have a negative pregnancy test at enrollment.
12. If a subject has received more than three prior regimens of cytotoxic chemotherapy, or more than two biological or targeted therapies, or more than 3000 cGy to >25% of his or her bone marrow, the investigator must discuss with the sponsor regarding subject suitability prior to enrollment.
13. The subject has had no other diagnosis of malignancy (unless non-melanoma skin cancer, in situ carcinoma of the cervix, or a malignancy diagnosed ≥5 years ago, and has had no evidence of disease for 5 years prior to screening for this study).

Exclusion Criteria:

1. The subject has received systemic anticancer therapy (eg, chemotherapy, biologic therapy, targeted therapy, cytokines, or hormones) within 14 days before the first dose of study drug.
2. The subject has received radiation to >25% of his or her bone marrow within 30 days of XL999 treatment.
3. The subject has not recovered to Grade ≤1 from adverse events (AEs) due to investigational or other agents administered more than 14 days prior to study enrollment.
4. The subject has history of or known brain metastases, current spinal cord compression, or carcinomatous meningitis.
5. The subject is known to be positive for the human immunodeficiency virus (HIV).
6. The subject has uncontrolled and/or intercurrent illness including but not limited to the following:

   1. Cardiac:

      * Left ventricular ejection fraction (LVEF) assessed by 99mTc multiple-gated acquisition scan (MUGA) is below the institution's lower limit of normal (LLN) at screening. If regional wall motion abnormalities are noted on the MUGA, cardiology consultation should be performed prior to enrollment.
      * History of pulmonary hypertension.
      * History of congestive heart failure (CHF) (New York Heart Association [NYHA] Class II, III, or IV).
      * Active or unstable ischemic disease, including angina pectoris, myocardial infarction, coronary artery bypass grafting (CABG) within the past 12 months.
      * Electrocardiogram (ECG) showing signs of ischemia or myocardial, valvular, or coronary artery disease unless deemed clinically insignificant by a cardiologist.
      * Onset of any changes between the screening ECG and pre-dose ECG unless deemed clinically insignificant by a cardiologist.
      * ECG abnormalities that could cause interpretation difficulties after XL999 administration (eg, left bundle branch block [LBBB], atrial fibrillation, A-V blocks, pacemakers, digoxin).
   2. Vascular:

      * Blood pressure >150/90 mm Hg despite antihypertensive therapy with two medications.
      * Cerebrovascular accident, transient ischemic attack, or evidence of active peripheral vascular disease within 12 months prior to study enrollment.
   3. Hematologic:

      * National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 Grade ≥3 hemorrhage within 30 days of study enrollment.
      * Evidence of bleeding diathesis or coagulopathy.
      * Requirement for therapeutic anticoagulation. Patients receiving anticoagulants (eg, warfarin, heparin) will be excluded if international normalized ratio >1.5 or partial thromboplastin time (PTT) >1.5× the institution's ULN.
   4. Recent surgical procedures:

      * Major surgery or open biopsy within 30 days of starting treatment with XL999.
      * Anticipation of major surgical procedure during the study.
   5. Wound healing problems:

      * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 30 days prior to treatment.
      * Serious, non-healing wound, ulcer, or bone fracture.
   6. Psychiatric illness that would limit compliance with study requirements.
7. The subject is pregnant or breastfeeding.
8. The subject has a known allergy or hypersensitivity to components of the XL999 formulation.
9. The subject is unable or unwilling to abide by the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, and maximum tolerated dose of XL999 administered weekly as a 4-hour intravenous infusion | Inclusion until 30 days post last treatment

SECONDARY OUTCOMES:
Plasma pharmacokinetics of XL999 administered weekly as a 4-hour intravenous infusion | At various time points during the 4 week Treatment Period and the Treatment Extension Period

CONTACTS AND LOCATIONS:
Overall Officials: Lynne A. Bui, MD, Study Director — Exelixis
Locations (5):
- United States (5):
  - UCLA Medical Center, Los Angeles, California
  - Peachtree Hematology Oncology Consultants, Atlanta, Georgia
  - Wayne State University, Karmanos Cancer Institute, Detroit, Michigan
  - Hematology-Oncology Associates of Rockland, Nyack, New York
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas